CLINICAL TRIAL: NCT02509624
Title: A Phase 1, Open-Label, Parallel-Group, Single Dose Study to Evaluate the Pharmacokinetics of GS-4997 in Subjects With Normal and Impaired Hepatic Function
Brief Title: Study to Evaluate the Pharmacokinetics of Selonsertib in Participants With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-223-1018; 2015-002444-14 (EudraCT Number)
Record Dates: First submitted 2015-07-16; First posted 2015-07-28 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — selonsertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate hepatic impairment (Cohort 1) (Experimental): Participants with moderate hepatic impairment and matched healthy controls will receive a single dose of selonsertib on Day 1.
  Interventions: Drug: Selonsertib
- Severe hepatic impairment (Cohort 2) (Experimental): Participants with severe hepatic impairment and matched healthy controls will receive a single dose of selonsertib on Day 1.
  Interventions: Drug: Selonsertib
- Mild hepatic impairment (Cohort 3) (Experimental): Participants with mild hepatic impairment and matched healthy controls will receive a single dose of selonsertib on Day 1.
  Interventions: Drug: Selonsertib

INTERVENTIONS:
Drug: Selonsertib — 6 mg tablets administered orally in fed state
  Other Names: GS-4997

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of selonsertib in participants with impaired hepatic function relative to matched, healthy controls.

ELIGIBILITY:
Key Inclusion Criteria:

All participants:

* Body mass index (BMI) from 18 to 40 kg/m^2, inclusive at study screening
* Creatinine clearance (CrCl) ≥ 60 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at screening

Participants with impaired hepatic function:

* Aside from hepatic insufficiency, participants must be sufficiently healthy for study participation based upon screening evaluations.
* Must have diagnosis of chronic (> 6 months), stable hepatic impairment with no clinically significant change in hepatic status within the 3 months (90 days) prior to study drug administration (Day 1).
* Participants with severe hepatic impairment must have a score on the Child-Pugh-Turcotte scale of 10-15 at screening.
* Participants with moderate hepatic impairment must have a score on the Child-Pugh-Turcotte scale of 7-9 at screening.
* Participants with mild hepatic impairment must have a score on the Child-Pugh-Turcotte scale of 5-6 at screening.

Healthy participants (matched control):

* Must be in good health based upon screening evaluations.

Key Exclusion Criteria:

All participants:

* Pregnant or lactating females
* Have received any investigational compound or device within 30 days prior to study dosing
* Current alcohol or substance abuse
* A positive test result for human immunodeficiency virus (HIV-1/2) antibody
* Have poor venous access that limits phlebotomy
* Have been treated with systemic steroids, anti-HIV agents, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to screening or expected to receive these agents during the study (eg, corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies) that would be contraindicated for other exclusion criteria.
* Significant serious skin disease, such as but not limited to rash, food allergy, eczema, psoriasis, or urticaria
* Significant drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
* Unstable cardiac disease, including history of myocardial infarction within 1 year of screening, recurrent episodes of ventricular tachycardia despite appropriate medical therapy, decompensated congestive heart failure, or dilated cardiomyopathy with left ventricular ejection fraction < 40%, or a family history of Long QT Syndrome, or unexplained death in an otherwise healthy participants between the ages of 1 and 30 years.
* Syncope, palpitations, or unexplained dizziness
* Implanted defibrillator or pacemaker
* Severe peptic ulcer disease, severe gastroesophageal reflux disease, or other severe gastric acid hypersecretory conditions
* Medical or surgical treatment that permanently alters gastric absorption (eg, gastric or intestinal surgery). A history of cholecystectomy is not exclusionary.
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation.
* Currently registered on an organ transplantation list.
* History of bleeding from esophageal varices within 90 days prior to Admission (Day -1).
* Use of strong cytochrome P3A4 (CYP3A4) inhibitors (eg, indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, suboxone, telithromycin, atazanavir) and strong CYP3A4 inducers (eg, carbamazepine, rifampin, phenytoin and St. John's wort), within 28 days prior to study drug administration (Day 1).
* Consumption of grapefruit juice, grapefruits, and Seville orange juice within 2 weeks prior to study drug administration (Day 1).
* Recent significant changes in the use of nicotine or nicotine containing products

Participants with impaired hepatic function:

* Aside from hepatic insufficiency, serious or active medical or psychiatric illness that, in the opinion of the investigator, would interfere with treatment, assessment, or compliance with the protocol.
* Chronic hepatitis B virus (HBV) infection, defined as a positive test for hepatitis B surface antigen (HBsAg), unless the participant has been treated with a nucleos(t)ide analog (eg, tenofovir or entecavir) for at least 6 months and the HBV deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR) assay has been persistently undetectable for at least 6 months.
* Positive test for drugs of abuse, including alcohol at screening or on Day -1/check-in, with the exception of opioids and tetrahydrocannabinol (THC, marijuana) under prescription and investigator verification for pain management. Participants who screen positive for benzodiazepines may be allowed if prescribed under the care of a physician and after review by investigator and Sponsor.
* Requires paracentesis > 1 time per month.
* Participants with hepatic impairment with co-morbid diseases not associated with hepatic impairment requiring medication(s) must be taking the medication(s) without a change in dose for > 3 months prior to screening.
* Changes in concomitant medications or dosage used to treat symptoms of hepatic impairment or associated co-morbid conditions that could lead to clinically significant changes in medical conditions during the course of the study that would affect the ability to interpret potential drug-drug interactions within 28 days prior to dosing.

Healthy participants (matched control):

* A positive test result for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (anti-HBc)
* Positive test for drugs of abuse, including alcohol at screening or on Day -1/check-in.
* Have any serious or active medical or psychiatric illness (including depression) which, in the opinion of the investigator, would interfere with treatment, assessment, or compliance with the protocol.
* History of liver disease.
* Have taken any prescription medications or over-the-counter medications including herbal products within 28 days of commencing study drug dosing with the exception of vitamins, acetaminophen, ibuprofen, and hormonal contraceptive medications.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Denver, Colorado
  - Miami, Florida
  - Orlando, Florida
  - Minneapolis, Minnesota
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 17 August 2015. The last study visit occurred on 15 December 2015.
Pre-assignment Details: 107 participants were screened. In the control groups (normal hepatic function), each participant was matched for age, gender, race, and body mass index with a participant in the hepatic impairment group. 22 total unique participants with normal hepatic function were enrolled in Cohorts 1, 2, and 3. 3 participants served as matched control in both Cohort 1 and 2. 1 participant served as a matched control in both Cohort 1 and 3. 4 participants served as matched control in both Cohort 2 and 3.
Groups:
- Cohort 1: Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
- Cohort 2: Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
- Cohort 3: Mild Hepatic Impairment: Participants with mild hepatic impairment received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
- Healthy Control: Matched normal hepatic function participants received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Healthy Control
Started | 10 | 10 | 10 | 22
Completed | 10 | 10 | 10 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Healthy Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 22 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (5.0) | 54 (5.8) | 53 (10.4) | 53 (8.4) | 54 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 5 | 13
  Male | 8 | 7 | 7 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 4 | 12 | 27
  Not Hispanic or Latino | 7 | 2 | 6 | 10 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 7 | 10
  White | 7 | 10 | 9 | 14 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCinf of Selonsertib and Its Metabolite GS-607509
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: 0 (predose), 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1. Additional PK samples were collected at the Day 10 and 14 follow-up visits approximately the same time as the Day 1 predose sample.
Population: PK Analysis Set included all enrolled participants who received at least 1 dose of selonsertib and had at least 1 evaluable PK concentration data value reported by the PK laboratory for the respective analytes. 3 participants served as matched control in both Cohort 1 and 2. 1 participant served as a matched control in both Cohort 1 and 3. 4 participants served as matched control in both Cohort 2 and 3.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Matched Healthy Control for Cohort 1: Matched normal hepatic function participants to moderate hepatic impairment received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
- Matched Healthy Control for Cohort 2: Matched normal hepatic function participants to severe hepatic impairment received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
- Matched Healthy Control for Cohort 3: Matched normal hepatic function participants to mild hepatic impairment received a single oral dose of selonsertib 6 mg (1 × 6 mg tablet) in fed state on Day 1.
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Matched Healthy Control for Cohort 1 | Matched Healthy Control for Cohort 2 | Matched Healthy Control for Cohort 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
hr*ng/mL
  AUCinf of Selonsertib | 3316.1 (1734.11) | 3266.7 (766.39) | 2962.1 (901.12) | 2835.3 (499.58) | 2277.9 (490.96) | 2711.6 (919.83)
  AUCinf of GS-607509 | 5941.8 (2286.80) | 5711.2 (3401.94) | 10203.6 (8689.39) | 9993.3 (4599.91) | 9603.4 (8057.84) | 9846.6 (8954.40)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Hepatic Impairment vs Matched Healthy Control for Cohort 1; AUCinf of selonsertib; Test type: Other; %Geometric least-square mean(GLSM) ratio = 105.08, 90% CI 2-sided [77.08 to 143.23]
Statistical Analysis 2: Comparison: Cohort 2: Severe Hepatic Impairment vs Matched Healthy Control for Cohort 2; AUCinf of selonsertib; Test type: Other; % GLSM ratio = 142.65, 90% CI 2-sided [120.52 to 168.84]
Statistical Analysis 3: Comparison: Cohort 3: Mild Hepatic Impairment vs Matched Healthy Control for Cohort 3; AUCinf of selonsertib; Test type: Other; % GLSM ratio = 110.55, 90% CI 2-sided [86.99 to 140.49]
Statistical Analysis 4: Comparison: Cohort 1: Moderate Hepatic Impairment vs Matched Healthy Control for Cohort 1; AUCinf of GS-607509; Test type: Other; % GLSM ratio = 62.05, 90% CI 2-sided [43.84 to 87.81]
Statistical Analysis 5: Comparison: Cohort 2: Severe Hepatic Impairment vs Matched Healthy Control for Cohort 2; AUCinf of GS-607509; Test type: Other; % GLSM ratio = 66.44, 90% CI 2-sided [36.72 to 120.21]
Statistical Analysis 6: Comparison: Cohort 3: Mild Hepatic Impairment vs Matched Healthy Control for Cohort 3; AUCinf of GS-607509; Test type: Other; % GLSM ratio = 103.46, 90% CI 2-sided [51.75 to 206.83]

2. Primary Outcome: PK Parameter: AUClast of Selonsertib and Its Metabolite GS-607509
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed. 3 participants served as matched control in both Cohort 1 and 2. 1 participant served as a matched control in both Cohort 1 and 3. 4 participants served as matched control in both Cohort 2 and 3.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Matched Healthy Control for Cohort 1 | Matched Healthy Control for Cohort 2 | Matched Healthy Control for Cohort 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
hr*ng/mL
  AUClast of Selonsertib | 2964.1 (1493.69) | 3032.7 (728.55) | 2790.8 (847.18) | 2679.9 (486.23) | 2129.7 (493.83) | 2530.9 (902.55)
  AUClast of GS-607509 | 5405.2 (2211.86) | 4868.0 (3072.43) | 8475.8 (7165.86) | 9117.6 (4127.22) | 8157.5 (6019.61) | 8326.5 (6604.26)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Hepatic Impairment vs Matched Healthy Control for Cohort 1; AUClast of selonsertib; Test type: Other; % GLSM ratio = 99.87, 90% CI 2-sided [73.38 to 135.92]
Statistical Analysis 2: Comparison: Cohort 2: Severe Hepatic Impairment vs Matched Healthy Control for Cohort 2; AUClast of selonsertib; Test type: Other; % GLSM ratio = 141.75, 90% CI 2-sided [118.50 to 169.55]
Statistical Analysis 3: Comparison: Cohort 3: Mild Hepatic Impairment vs Matched Healthy Control for Cohort 3; AUClast of selonsertib; Test type: Other; % GLSM ratio = 112.24, 90% CI 2-sided [87.69 to 143.65]
Statistical Analysis 4: Comparison: Cohort 1: Moderate Hepatic Impairment vs Matched Healthy Control for Cohort 1; AUClast of GS-607509; Test type: Other; % GLSM ratio = 61.20, 90% CI 2-sided [43.06 to 86.98]
Statistical Analysis 5: Comparison: Cohort 2: Severe Hepatic Impairment vs Matched Healthy Control for Cohort 2; AUClast of GS-607509; Test type: Other; % GLSM ratio = 61.07, 90% CI 2-sided [33.62 to 110.91]
Statistical Analysis 6: Comparison: Cohort 3: Mild Hepatic Impairment vs Matched Healthy Control for Cohort 3; AUClast of GS-607509; Test type: Other; % GLSM ratio = 96.13, 90% CI 2-sided [48.47 to 190.67]

3. Primary Outcome: PK Parameter: Cmax of Selonsertib and Its Metabolite GS-607509
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Matched Healthy Control for Cohort 1 | Matched Healthy Control for Cohort 2 | Matched Healthy Control for Cohort 3
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
ng/mL
  Cmax of Selonsertib | 93.7 (20.66) | 82.4 (10.63) | 110.6 (24.77) | 105.4 (22.13) | 91.9 (22.01) | 110.3 (23.40)
  Cmax of GS-607509 | 44.1 (15.01) | 31.2 (15.34) | 63.5 (31.42) | 62.3 (23.44) | 63.2 (27.03) | 64.2 (21.99)
Statistical Analysis 1: Comparison: Cohort 1: Moderate Hepatic Impairment vs Matched Healthy Control for Cohort 1; Cmax of selonsertib; Test type: Other; % GLSM ratio = 88.68, 90% CI 2-sided [74.83 to 105.10]
Statistical Analysis 2: Comparison: Cohort 2: Severe Hepatic Impairment vs Matched Healthy Control for Cohort 2; Cmax of selonsertib; Test type: Other; % GLSM ratio = 91.16, 90% CI 2-sided [78.76 to 105.52]
Statistical Analysis 3: Comparison: Cohort 3: Mild Hepatic Impairment vs Matched Healthy Control for Cohort 3; Cmax of selonsertib; Test type: Other; % GLSM ratio = 100.19, 90% CI 2-sided [83.73 to 119.88]
Statistical Analysis 4: Comparison: Cohort 1: Moderate Hepatic Impairment vs Matched Healthy Control for Cohort 1; Cmax of GS-607509; Test type: Other; % GLSM ratio = 71.44, 90% CI 2-sided [54.58 to 93.50]
Statistical Analysis 5: Comparison: Cohort 2: Severe Hepatic Impairment vs Matched Healthy Control for Cohort 2; Cmax of GS-607509; Test type: Other; % GLSM ratio = 46.92, 90% CI 2-sided [32.59 to 67.54]
Statistical Analysis 6: Comparison: Cohort 3: Mild Hepatic Impairment vs Matched Healthy Control for Cohort 3; Cmax of GS-607509; Test type: Other; % GLSM ratio = 93.93, 90% CI 2-sided [67.60 to 130.50]

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Study Drug-related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant which did not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-emergent AEs were defined as events that met one of the following criteria: 1) Any AEs with an onset date of on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug; or 2) Any AEs leading to premature discontinuation of study drug.
Time Frame: Day 1 plus 30 days
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10 | 10 | 22
percentage of participants | 20.0 | 0 | 10.0 | 13.6

5. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-Emergent and Grade ≥ 3 Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increased at least 1 toxicity grade from predose at any postdose visit, up to and including the date of last dose of study drug plus 30 days for participants who permanently discontinued study drug. If the relevant baseline laboratory value was missing, then any abnormality of at least Grade 1 observed within the time frame specified above was considered treatment-emergent. Severity grades were defined based on modified Common Terminology Criteria for Adverse Events (CTCAE) Laboratory Abnormality and Adverse Event Severity Grading, where 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Day 1 plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10 | 10 | 22
percentage of participants
  Any Treatment-Emergent Laboratory Abnormalities | 90.0 | 90.0 | 70.0 | 59.1
  Grade ≥ 3 Laboratory Abnormalities | 20.0 | 40.0 | 10.0 | 4.5

ADVERSE EVENTS:
Time Frame: Day 1 plus 30 days
Description: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: Moderate Hepatic Impairment | Cohort 2: Severe Hepatic Impairment | Cohort 3: Mild Hepatic Impairment | Healthy Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 3/10 | 0/10 | 2/10 | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Moderate Hepatic Impairment (N=10) | Cohort 2: Severe Hepatic Impairment (N=10) | Cohort 3: Mild Hepatic Impairment (N=10) | Healthy Control (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years